CLINICAL TRIAL: NCT03722303
Title: Lipografting Versus Steroid Injections for Treatment of Primary Mild to Moderate Carpal Tunnel Syndrome
Brief Title: Lipografting Versus Steroid Injections for Treatment of Carpal Tunnel Syndrome
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Columbia University (Other)
Collaborators: Orthopaedic Scientific Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AAAK4700
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal; tunnel; injection; steroid; lipografting; numbness; tingling; median nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome; Hypesthesia; Paresthesia | interventions — CD36 Antigens; Steroids; Cortisone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid Injection (Active Comparator): Subjects with CTS will receive steroid injection.
  Interventions: Drug: Steroid Injection
- Fat Injection (Experimental): Subjects with CTS will receive fat injection.
  Interventions: Other: Fat Injection

INTERVENTIONS:
Other: Fat Injection — Used by plastic surgeons, lipografting injects autologous fat to correct contour deformities. Plastic surgeons have witnessed the regenerative properties of fat transfer, and these clinical manifestations have fostered numerous studies defining fat as a rich source of pluripotent stem cells with the potential for reducing scar formation, bringing neo-angiogenesis, and providing a barrier against scar adhesions. This study applies the regenerative properties of autologous fat transfer to treat mild to moderate carpal tunnel syndrome in comparison to the current standard of care, corticosteroid treatment. Ideally, fat transfer would prevent scar formation and aid in nerve excursion along the canal, while the neoangiogenic and regenerative growth factors stimulate nerve regeneration.
  Other Names: Fat Transfer
  Arms: Fat Injection
Drug: Steroid Injection — Standard of care non-operative treatment for the treatment of Carpal Tunnel Syndrome
  Other Names: Cortisone Injection
  Arms: Steroid Injection

SUMMARY:
This study applies the regenerative properties of autologous fat transfer to treat mild to moderate carpal tunnel syndrome in comparison to the current standard of care, corticosteroid treatment. The investigators hypothesize the fat transfer would prevent scar formation and aid in nerve excursion along the canal (while the neoangiogenic and regenerative growth factors could stimulate nerve regeneration) better than the standard of care treatment.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy affecting up to 13% of Americans; CTS is caused by compression of the median nerve in the carpal tunnel leading to nerve ischemia and symptoms of numbness, pain, and tingling. Treatment options depend on the severity of symptoms and range from noninvasive options (most commonly, steroid injections) to definitive surgical release of the compressed median nerve. Both non-invasive techniques and surgical intervention have their shortcomings; thus a novel approach for CTS treatment may be indicated.

Lipografting is an established, validated, and widely used technique of plastic surgeons that injects autologous fat to correct contour deformities. From observing these reconstructions, plastic surgeons have witnessed the regenerative properties of fat transfer, specifically delaying the affects of chronic radio-dermatitis. These clinical manifestations have fostered numerous studies defining fat as a rich source of pluripotent stem cells with the potential for reducing scar formation, bringing neo-angiogenesis, and providing a barrier against scar adhesions This study applies the regenerative properties of autologous fat transfer to treat mild to moderate carpal tunnel syndrome in comparison to the current standard of care, corticosteroid treatment. Ideally, the fat transfer would prevent scar formation and aid in nerve excursion along the canal, while the neoangiogenic and regenerative growth factors could stimulate nerve regeneration.

ELIGIBILITY:
Inclusion Criteria:

* primary mild to moderate carpal tunnel syndrome (CTS)
* report symptoms longer than 6 months
* night pain
* weakness
* sensory deficits
* fluent English-speaking adult (>18)

Exclusion Criteria:

* <18 years old
* Non-english speaking
* injection in past 6 months
* previous hand surgery
* previous hand trauma (fracture or dislocation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Functional Outcome Score | Up to 1 year post-treatment
  This score will be determined by Quick-Disabilities of the Arm, Shoulder and Hand (QuickDASH), which is a validated tool/survey for measuring upper extremity disability. The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (4 items, scored 1-5). These raw scores are used to calculate a score out of 100, with a higher score indicating greater disability.

SECONDARY OUTCOMES:
Score on the Michigan Hand Questionnaire (MHQ) | Up to 1 year post-treatment
  The MHQ is hand-specific outcomes instrument that measures outcomes of patients with conditions of, or injury to, the hand or wrist. In the pain scale, high scores indicate greater pain, while in the other five scales, high scores denote better hand performance.
Score on the Brigham Women's Carpal Tunnel Questionnaire | Up to 1 year post-treatment
  Brigham Women's Carpal Tunnel Questionnaire is a validated tool for measuring severity of symptoms for carpal tunnel syndrome. The questionnaire is self-administered, with each item scored from 1 to 5 (where 1 indicates no symptoms or no functional difficulty, and 5 indicates maximum symptoms or an inability to perform the functional task).

CONTACTS AND LOCATIONS:
Overall Officials: Melvin P Rosenwasser, MD, Principal Investigator — Department of Orthopaedic Surgery at Columbia University Medical Center
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LeBlanc KE, Cestia W. Carpal tunnel syndrome. Am Fam Physician. 2011 Apr 15;83(8):952-8. PMID 21524035
- [Background] Marshall S, Tardif G, Ashworth N. Local corticosteroid injection for carpal tunnel syndrome. Cochrane Database Syst Rev. 2007 Apr 18;2007(2):CD001554. doi: 10.1002/14651858.CD001554.pub2. PMID 17443508
- [Background] Gutowski KA; ASPS Fat Graft Task Force. Current applications and safety of autologous fat grafts: a report of the ASPS fat graft task force. Plast Reconstr Surg. 2009 Jul;124(1):272-280. doi: 10.1097/PRS.0b013e3181a09506. PMID 19346997
- [Background] Ibrahim I, Khan WS, Goddard N, Smitham P. Carpal tunnel syndrome: a review of the recent literature. Open Orthop J. 2012;6:69-76. doi: 10.2174/1874325001206010069. Epub 2012 Feb 23. PMID 22470412